CLINICAL TRIAL: NCT03275766
Title: Effects of Transcranial Magnetic Stimulation on Motor Symptoms of Patients With Psychiatric Disorders
Brief Title: Transcranial Magnetic Stimulation (TMS) for Motor Symptoms in Psychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Principal Investigator, Sebastian Walther, Prof. Dr., Head of the outpatient clinic, University Hospital of Psychiatry, University of Bern
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SNCTP610
Record Dates: First submitted 2017-08-22; First posted 2017-09-08 (Actual); Results first posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Psychomotor Retardation; Psychomotor Slowing; Schizophrenia and Related Disorders; Major Depressive Disorder
MeSH Terms: conditions — Psychomotor Disorders; Schizophrenia; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DLPFC facilitatory (Active Comparator): repetitive transcranial magnetic stimulation (rTMS) of 15 Hz over left DLPFC
  usually effective in depression treatment, probably no specific effect on psychomotor slowing
  Interventions: Other: DLPFC facilitatory
- preSMA/SMA inhibitory (Experimental): repetitive transcranial magnetic stimulation (rTMS) of 1 Hz over preSMA/SMA
  should inhibit overactive premotor cortices
  Interventions: Other: SMA inhibitory
- preSMA/SMA facilitatory (Experimental): intermittend theta burst stimulation (iTBS) over preSMA/SMA
  should facilitate neural activity within premotor cortices
  Interventions: Other: SMA facilitatory
- sham TMS (Sham Comparator): sham rTMS with a placebo coil over occipital cortex
  should have no effect at all (no transcranial magnetic stimulation, only sound)
  Interventions: Other: sham TMS

INTERVENTIONS:
Other: DLPFC facilitatory — 15 Hz stimulation of left dorsolateral prefrontal cortex (DLPFC)(15 sessions/3weeks, 1500 stimuli per session, stimulation intensity 100% of the individual active motor threshold; in total 22500 stimuli
  Other Names: rTMS facilitatory DLPFC
  Arms: DLPFC facilitatory
Other: SMA inhibitory — 1 Hz stimulation of preSMA/SMA (15 sessions/3weeks, 1500 stimuli per session, stimulation intensity 100% of the individual active motor threshold; in total 22500 stimuli
  Other Names: rTMS inhibitory SMA
  Arms: preSMA/SMA inhibitory
Other: SMA facilitatory — Three pulses of stimulation at 50 Hz of preSMA/SMA, repeated every 200 ms. 2 s trains are repeated every 10 s for a total of 190 s (600 pulses, 200 seconds). intensity 80% of individual active motor threshold; in total 9000 stimuli
  Other Names: iTBS facilitatory SMA
  Arms: preSMA/SMA facilitatory
Other: sham TMS — Determination of active motor threshold and subsequent stimulation with the placebo coil, with the same sounds but without effects. 15 sessions in three weeks, duration of 20 mins per session
  Arms: sham TMS

SUMMARY:
Psychomotor slowing may occur in major psychiatric disorders, such as major depressive disorders or schizophrenia spectrum disorders. It refers to slowing of fine motor skills, motor planning and gross motor behavior. In major depression and schizophrenia, psychomotor slowing is associated with alterations of premotor cortex, dorsolateral prefrontal cortex and basal ganglia. This randomized, sham-controlled, prospective trial will test, whether 15 sessions of repetitive transcranial magnetic stimulation (rTMS) may ameliorate psychomotor slowing in schizophrenia or major depression.

DETAILED DESCRIPTION:
Psychomotor slowing may occur in major psychiatric disorders, such as major depressive disorders or schizophrenia spectrum disorders. It refers to slowing of fine motor skills, motor planning and gross motor behavior. In major depression and schizophrenia, psychomotor slowing is associated with alterations of premotor cortex, dorsolateral prefrontal cortex and basal ganglia. This randomized, sham-controlled, prospective trial will test, whether 15 sessions of rTMS in 3 weeks may ameliorate psychomotor slowing in schizophrenia or major depression.

Eligible participants will be randomized to one of four arms:

ELIGIBILITY:
Inclusion Criteria:

* suffering from major depressive disorder or schizophrenia spectrum disorder according to DSM-5 criteria
* right handedness
* normal or corrected-to-normal vision and hearing

Exclusion Criteria:

* epilepsy
* history of severe head trauma
* current abuse of drugs or alcohol; past addiction to drugs or alcohol
* pregnancy
* incompatibility to cerebral MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Walther, MD, Principal Investigator — University of Bern, University Hospital of Psychiatry
Locations (1):
- University Hospital of Psychiatry, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DLPFC Facilitatory: repetitive transcranial magnetic stimulation (rTMS) of 15 Hz over left DLPFC
  usually effective in depression treatment, probably no specific effect on psychomotor slowing
  DLPFC facilitatory: 15 Hz stimulation of left dorsolateral prefrontal cortex (DLPFC)(15 sessions/3weeks, 1500 stimuli per session, stimulation intensity 100% of the individual active motor threshold; in total 22500 stimuli
- preSMA/SMA Inhibitory: repetitive transcranial magnetic stimulation (rTMS) of 1 Hz over preSMA/SMA
  should inhibit overactive premotor cortices
  SMA inhibitory: 1 Hz stimulation of preSMA/SMA (15 sessions/3weeks, 1500 stimuli per session, stimulation intensity 100% of the individual active motor threshold; in total 22500 stimuli
- preSMA/SMA Facilitatory: intermittend theta burst stimulation (iTBS) over preSMA/SMA
  should facilitate neural activity within premotor cortices
  SMA facilitatory: Three pulses of stimulation at 50 Hz of preSMA/SMA, repeated every 200 ms. 2 s trains are repeated every 10 s for a total of 190 s (600 pulses, 200 seconds). intensity 80% of individual active motor threshold; in total 9000 stimuli
- Sham TMS: sham rTMS with a placebo coil over occipital cortex
  should have no effect at all (no transcranial magnetic stimulation, only sound)
  sham TMS: Determination of active motor threshold and subsequent stimulation with the placebo coil, with the same sounds but without effects. 15 sessions in three weeks, duration of 20 mins per session
Period: Overall Study
Arm/Group | DLPFC Facilitatory | preSMA/SMA Inhibitory | preSMA/SMA Facilitatory | Sham TMS
Started | 12 | 12 | 11 | 10
Received Intervention | 9 | 11 | 10 | 9
Completed | 7 | 5 | 7 | 4
Not Completed | 5 | 7 | 4 | 6

BASELINE CHARACTERISTICS:
Population: one subject randomized withdrew consent before the baseline assessments
Groups:
- Total: Total of all reporting groups
Arm/Group | DLPFC Facilitatory | preSMA/SMA Inhibitory | preSMA/SMA Facilitatory | Sham TMS | Total
Number analyzed (Participants) | 12 | 11 | 11 | 10 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 11 | 10 | 44
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (15.2) | 38.0 (15.6) | 34.2 (14.0) | 41.2 (15.3) | 39.5 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 3 | 13
  Male | 10 | 8 | 6 | 7 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 12 | 11 | 11 | 10 | 44
Diagnosis [Number; unit: participants]
  major depression | 5 | 5 | 5 | 4 | 19
  schizophrenia | 7 | 6 | 6 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders at Week 3
Description: Number of participants with >30% reduction from baseline in the Salpetriere Retardation Rating Scale, last observation carried forward method applied
Time Frame: week 3
Measure: Number; unit: responders
Arm/Group | DLPFC Facilitatory | preSMA/SMA Inhibitory | preSMA/SMA Facilitatory | Sham TMS
Number analyzed (Participants) | 12 | 11 | 11 | 10
responders | 4 | 9 | 0 | 3

2. Secondary Outcome: Change in Salpetriere Retardation Rating Scale Total Score From Baseline to Week 3
Description: observer based rating scale of the severity of psychomotor slowing, assessment blind to intervention Scores may range from 0 - 60, higher scores indicate worse outcome
Time Frame: week 3
Reporting Status: Not Posted

3. Secondary Outcome: Change in Activity Level From Baseline to Week 3
Description: actigraphically (wrist of the non-dominant arm) assessed motor activity during the wake periods of one day, given in counts/h
Time Frame: week 3
Reporting Status: Not Posted

4. Secondary Outcome: Change in Catatonia Severity From Baseline to Week 3
Description: observer based rating of catatonia severity with the Bush Francis Catatonia Rating Scale, assessment blind to intervention
Time Frame: week 3
Reporting Status: Not Posted

5. Secondary Outcome: Change in Fingertapping Score From Baseline to Week 3
Description: Fingertapping test with the dominant and nondominant index finger for 10 sec, video-taped and blind assessment
Time Frame: week 3
Reporting Status: Not Posted

6. Secondary Outcome: Change in Coin Rotation From Baseline to Week 3
Description: test of manual dexterity in both hands, rotation of a specified coin for 10 seconds, video-taped and blinded evaluation
Time Frame: week 3
Reporting Status: Not Posted

7. Secondary Outcome: Change in Hand Gesture Performance From Baseline to Week 3
Description: videotaped performance of hand gestures according to the Test of Upper Limb Apraxia (TULIA), blind evaluation and rating
Time Frame: week 3
Reporting Status: Not Posted

8. Secondary Outcome: Change in SANS Total Score From Baseline to Week 3
Description: scale for the assessment of negative symptoms, applies to schizophrenia spectrum disorder patients, assessment blind to intervention
Time Frame: week 3
Reporting Status: Not Posted

9. Secondary Outcome: Change From HAMD Total Score From Baseline to Week 3
Description: Hamilton Rating Scale for Depression, 21-item version, applies to depression patients, assessment blind to intervention
Time Frame: week 3
Reporting Status: Not Posted

10. Secondary Outcome: Change in CAINS Total Score From Baseline to Week 3
Description: the clinical assessment interview for negative symptoms, assessment blind to intervention
Time Frame: week 3
Reporting Status: Not Posted

11. Secondary Outcome: Change in PANSS Total and Subscores From Baseline to Week 3
Description: the positive and negative syndrome scale, interview to assess severity of schizophrenia symptoms, applies to schizophrenia spectrum disorder patients, assessment blind to intervention
Time Frame: week 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data was collected during and after the daily rTMS sessions, inquiry covered the total three weeks of the trial
Description: inquiry with open questions
Arm/Group | DLPFC Facilitatory | preSMA/SMA Inhibitory | preSMA/SMA Facilitatory | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 1/12 | 1/11 | 0/11 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLPFC Facilitatory (N=12) | preSMA/SMA Inhibitory (N=11) | preSMA/SMA Facilitatory (N=11) | Sham TMS (N=10)
Deterioration of psychiatric disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — one patient experienced a deterioration of the underlying psychiatric disorder (major depression), which required short term hospitalization. The intervention was stopped. The problem resolved and the patient was discharged from the hospital.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DLPFC Facilitatory (N=12) | preSMA/SMA Inhibitory (N=11) | preSMA/SMA Facilitatory (N=11) | Sham TMS (N=10)
mild nausea (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
altered visual perception (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03275766/Prot_SAP_000.pdf